CLINICAL TRIAL: NCT07205445
Title: Tensi+ European Registry
Status: Recruiting | Type: Observational
Sponsor: Stimuli Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-A01420-47
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Overactive Bladder
Keywords: Urology; TENS; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tensi+ — Tensi+ (Stimuli Technology, Boulogne Billancourt, France) is a newly released, medical transcutaneous-posterior tibial nerve stimulation (TC-pTNS) device marketed for overactive bladder (OAB) management.

SUMMARY:
Tensi+ (Stimuli Technology, Boulogne Billancourt, France) is a newly released, medical transcutaneous-posterior tibial nerve stimulation (TC-pTNS) device marketed for overactive bladder (OAB) management. Preliminary studies have shown a favorable safety and efficacy profile. The goal of the present registry is to collect data among an important number of patients to assess the efficacy, safety and potential predictive factors of success in a current clinical setting over a total period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients suffering from idiopathic or neurological overactive bladder

Exclusion Criteria:

* Patients with pacemaker, defibrillator, or any other electronic implant;
* Patients with metal implant near the stimulation area;
* Pregnant women;
* People suffering from ankle joint problems, swollen ankles or a dermatological condition or damaged skin in the area where the electrodes are to be placed;
* Patient with cognitive impairment;
* Inability to complete a voiding diary;
* No social security cover (for applicable countries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years Overactive bladder symptoms
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Subjective improvement | 3 and 12 months
  The Patient Global Impression of Improvement (PGI-I) uses a 7-point scale, where post-treatment condition is rated as follows:
  1. = Very much better
  2. = Much better
  3. = A little better
  4. = No change
  5. = A little worse
  6. = Much worse
  7. = Very much worse.
  For analysis, patients with a PGI-I score of 1, 2, or 3 are typically considered responders, reflecting meaningful improvement.

SECONDARY OUTCOMES:
Patient-reported Outcomes Measures (PROMs) | 0; 3 and 12 months
  Urinary symptoms by filling up International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) which is a questionnaire intended to assess female storage, voiding and incontinence symptoms. Lower scores are typically associated with reduced symptom severity.
Patient-reported Outcomes Measures (PROMs) | 0; 3 and 12 months
  Urinary symptoms by filling up International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) which is a questionnaire intended to assess male storage, voiding and incontinence symptoms. Lower scores are typically associated with reduced symptom severity.
Quality of life measures | 0; 3 and 12 months
  By filling up International Consultation on Incontinence Questionnaire - OAB quality of life (ICIQ-OABqol) which is a questionnaire evaluating quality of life in patients with overactive bladder. Lower scores are typically associated with improved quality of life.

OTHER OUTCOMES:
Patient-reported Outcomes Measures (PROMs) | 0; 3 and 12 months
  By filling up International Consultation on Incontinence Questionnaire - Bowel (ICIQ-B) which is a questionnaire for evaluating symptoms of anal incontinence. Lower scores are typically associated with reduced symptom severity.
Evaluation of voiding frequency | 0; 3 and 12 months
  Evaluation of daytime voiding frequency averaged over three days from bladder diary entries
Evaluation of urgency | 0; 3 and 12 months
  Evaluation of daily urgency episodes averaged over three days from bladder diary entries
Evaluation of nocturia | 0; 3 and 12 months
  Evaluation of nocturia episodes averaged over three days from bladder diary entries
Evaluation of urgency urinary incontinence | 0; 3 and 12 months
  Evaluation of urgency urinary incontinence episodes averaged over three days from bladder diary entries
Evaluation of adverse events | 3 and 12 months
  Patients will be asked whether they experienced any adverse events during treatment. Patient responses will be collected and described qualitatively, enabling the identification of the types of adverse events reported as well as the frequency of their occurrence.

CONTACTS AND LOCATIONS:
Locations (15):
- France (3):
  - HFME - Hospices Civils de Lyon, Bron
  - CHU de Rennes, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
- Italy (9):
  - Nuova Villa Esther, Avellino
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Hesperia Hospital, Modena
  - Santa Maria la Gruccia Hospital, Montevarchi
  - Policlinico Tor Vergata, Roma
  - Casa di Cura Villa Stuart, Roma
  - Villa Salaria Hospital, Roma
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Clinica Nuova Villa Claudia, Roma
- United Kingdom (3):
  - Bristol Urological Institute, Bristol
  - Addenbrooke's Hospital, Cambridge University Hospital Trust, Cambridge
  - University College Hospital London, London

IPD SHARING:
Plan to Share IPD: No